CLINICAL TRIAL: NCT05920863
Title: Lenvatinib Combined with Tislelizumab and TACE Applied As Neoadjuvant Regimen for the Patients of CNLC Stage IB and IIA Hepatocellular Carcinoma with High Risk of Recurrence: Study Protocol of a Monocenter, Single-arm, Open Label Clincal Trail
Brief Title: Lenvatinib Combined with Tislelizumab and TACE Applied As Neoadjuvant Regimen for the Patients of CNLC Stage IB and IIA Hepatocellular Carcinoma with High-risk Recurrence Factors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yuhua Zhang, MD, Vice director of Hepatobiliary and Pancreatic Surgery (Chair), Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230408
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma; Lenvatinib; Tislelizumab; TACE; Pharmorubicin; Oxaliplatin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open phase II clinical study
Masking Description: Prior to enrollment in the study, doctors asked and recorded the patient's medical history, and if eligible participants volunteered to participate in the study, they would sign informed consent.If they are not willing to participate in the study, we will do the usual treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): 1. TACE: pharmorubicin 30mg, oxaliplatin 50mg, cycle 4-5 week.
  2. Tislelizumab: 200mg, cycle 3 week.
  3. Lenvatinib: weight <60kg, 8mg/day; weight ≥60kg, 12mg/day.
  Interventions: Procedure: TACE; Drug: Tislelizumab, Lenvatinib

INTERVENTIONS:
Procedure: TACE — TACE: pharmorubicin 30mg, oxaliplatin 50mg, cycle 4-5 week.
Drug: Tislelizumab, Lenvatinib — Tislelizumab: 200mg, cycle 3 week. Lenvatinib: weight <60kg, 8mg/day; weight ≥60kg, 12mg/day.

SUMMARY:
This is a monocenter, single-arm, open-label study to evaluate the efficacy and safety of Lenvatinib combined with Tislelizumab and TACE applied as neoadjuvant regimen for the patients of CNLC stage IB and IIA hepatocellular carcinoma with high risk of recurrence Primary outcome: Major pathological response (MPR) Secondary outcomes: pathological complete response (pCR), R0 resection rate, objective response rate (ORR), disease control rate (DCR), treatment-related adverse events (TRAE)

DETAILED DESCRIPTION:
Surgical treatment is dominant in the treatment of liver cancer, however, its postoperative recurrence rate is high, and the recurrence and metastasis rate in 5 years is as high as 70%. In particular, surgical resection for some large hepatocellular carcinoma adjacent to large vessels or located in middle areas always induces narrow and even no surgical margin, which may increase the risk of postoperative recurrence and decrease the overall survival rate. Preoperative neoadjuvant therapy for resectable hepatocellular carcinoma with high risk of recurrence is still controversial nationally and internationally, none consensus have been reached about neoadjuvant therapy.

As a classical treatment for liver cancer, TACE can induce tumor ischemia and necrosis through the infusion of chemotherapy drugs and embolic materials into target areas. However, TACE as neoadjuvant therapy alone has no improvement in tumor recurrence-free survival time and overall survival rate. Lenvatinib is a multi-target tyrosine kinase inhibitor and inhibits neovascularization and lymphangiogenesis by targeting VEGF1-3 and FGFR. moreover, lenvatinib also has immunomodulatory effects. A number of studies have shown that a variety of combination therapies have been carried out on the basis of Lenvatinib, and exciting outcome has been achieved by combined therapy regimens, including local therapy combined with systemic therapy and multi-drugs systemic therapy.

Neoadjuvant therapy will performe on CNLC stage IB and Stage IIA HCC patients with high risk of recurrence (patients with narrow or no surgical margin and preoperative tumor marker AFP+PIVKA≥1600). MPR, pCR,1-year recurrence-free survival (RFS), and treatment-related adverse reactions (TRAE) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old (inclusive);
2. HCC is confirmed by preoperative pathological examination or meet the criterion of diagnosis and treatment norms of primary HCC issued by health commission, PRC. No prior systemic chemotherapy, immunotherapy, targeted therapy, or other anti-tumor treatments for HCC;
3. Patients with CNLC IB or IIA stage tumors before surgery and meeting the following conditions: radiological evaluation shows narrow or none surgical margins, and preoperative tumor markers AFP+PIVKA is greater than 1600.
4. ECOG score of 0 before the first administration of the study drug;
5. Child-Pugh scores is 5-6 points and liver function is grade A;
6. Expected survival time of at least 16 weeks;
7. Pre-administration organ function levels meet the requirements and are tolerant of surgery. The functional indicators of important organs meet the following requirements: hemoglobin ≥90g/L, neutrophil count ≥1.5×10⁹/L, platelet count ≥100×10⁹/L; aspartate aminotransferase or alanine aminotransferase ≤5 times the upper limit of normal (ULN), alkaline phosphatase ≤2.5 ULN, serum albumin ≥30g/L; serum creatinine <1.5 ULN; international normalized ratio (INR) ≤2 or prothrombin time (PT) within the upper limit of normal range ≤6 seconds; serum creatinine ≤1.5 ULN, creatinine clearance rate ≥60 mL/min.
8. Male and female participants of childbearing potential must agree to use effective contraception throughout the study period;
9. Sign an informed consent form and agree to provide previously stored tumor tissue specimens or fresh biopsy specimens of the tumor lesion.

Exclusion Criteria:

1. Pathologically diagnosed as non-hepatocellular carcinoma;
2. Previously received anti-tumor treatments such as chemotherapy, radiotherapy, radiofrequency ablation, intervention, targeted therapy, immunotherapy or surgical treatment for liver cancer (excluding previous non-tumor-related surgery or diagnostic biopsy);
3. CNLC stage is IA, IIB or worse.
4. Viral load limited to hepatitis B virus (HBV) DNA>2000 copies/ml, hepatitis C virus (HCV) RNA>1000;
5. Long-term steroid users who require long-term systemic steroid therapy (equivalent to >10 mg of prednisone per day) or any other form of immunosuppressive treatment;
6. Significant clinical bleeding or bleeding tendency within 3 months before enrollment or currently undergoing thrombolysis or anticoagulation treatment;
7. Complete intestinal obstruction and incomplete intestinal obstruction requiring treatment, but patients who have had obstruction relieved by fistula or stent placement can be enrolled;
8. Active severe clinical infection (> grade 2, NCI-CTCAE version 5.0), including active tuberculosis; history of active tuberculosis infection for more than 1 year before enrollment, not treated with regular anti-tuberculosis treatment or tuberculosis still in the active period; active known or suspected autoimmune disease;
9. Uncontrolled diabetes (fasting blood glucose ≥10 mmol/L), severe lung disease (such as acute pulmonary disease, pulmonary fibrosis that affects lung function, interstitial lung disease. Excluding recovered radiation pneumonitis);
10. Clinically significant cardiovascular disease; hypertension which cannot be well controlled by anti-hypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
11. Patients undergoing renal replacement therapy;
12. History of other malignant tumors within the past 5 years. Excluding cured basal cell carcinoma or cervical intraepithelial neoplasia;
13. Other patients who are expected to be unable to tolerate surgical treatment;
14. Patients who have had allergic reactions to any component of the study drug;
15. Presence of alcohol dependence, mental illness, pregnancy (or lactation) or other conditions that are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response | Up to 16 weeks
  Proportion of residual tumor ingredient lesser than 30% in the postoperative pathological result.

SECONDARY OUTCOMES:
Pathological complete response | Up to 16 weeks
  None residual tumor ingredient detected in the postoperative pathological result.
R0 resection rate | Up to 16 weeks
  The proportion of patients achieved a complete resection with negative margin.
Objective response rate (ORR) | Up to 4 cycle treatment (each cycle is 4 weeks), an average of 16 weeks.
  he proportion of participants with a documented, confirmed complete response or partial response per RECIST v1.1
disease control rate (DCR) | Up to 4 cycle treatment (each cycle is 4 weeks), an average of 16 weeks.
  The percentage of patients who have achieved either a complete response (CR), a partial response (PR), or stable disease (SD) after undergoing treatment for their cancer.
treatment-related adverse events (TRAE) | Up to 4 cycle treatment (each cycle is 4 weeks), an average of 16 weeks.
  Adverse event that occurs during or after treatment
Recurrence-free survival (RFS) | Up to 4 cycle treatment (each cycle is 4 weeks), an average of 16 weeks.
  The length of time after cancer treatment during which a patient remains free from any signs or symptoms of cancer recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- 1# Banshan East Rd. Zhejiang cancer hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No